CLINICAL TRIAL: NCT06827236
Title: A Phase I/II, Multi-site, Open-label, Two-part Trial to Evaluate the Efficacy, Safety, and Pharmacokinetics of BNT323 in Combination With BNT327 in Participants With Advanced Breast Cancer
Brief Title: A Clinical Study to Find the Optimal Dose of an Investigational Treatment Called BNT323 When Used in Combination With Another Investigational Treatment, BNT327, and to Test if That Combination Treatment is Safe and Beneficial for Patients With Advanced Breast Cancer
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: BioNTech SE (Industry)
Collaborators: DualityBio Inc. (Industry); Biotheus Inc. (Industry); BioNTech (Shanghai) Pharmaceuticals Co., Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BNT323-03; 2024-517979-20-00 (EU CTIS Number); 1011776 (Other: IRAS number)
Record Dates: First submitted 2025-02-10; First posted 2025-02-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Locally Advanced Breast Cancer; Unresectable Breast Carcinoma; Metastatic Breast Cancer
Keywords: Breast Cancer (BC); Human epidermal growth factor receptor 2 (HER2); IHC scores 0, 1+, 2+, and 3+; Antibody drug conjugate (ADC); Programmed Death-1 (PD-1); Programmed Death Ligand-1 (PD-L1); Programmed Death-1 monoclonal antibodies; Anti vascular endothelial growth factor-A (anti-VEGF-A)
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Part1 - BNT323 + BNT327 combination therapy (Experimental): Escalating dose levels (DLs) of BNT323 and BNT327 to define RP2D. Six DLs are planned, i.e., DL0-1, DL1-1, DL2-1, DL0-0, DL1-0, DL2-0, a combination of three different DLs for BNT323 (DL0, DL1, and DL2) and two DLs for BNT327 (DL0 and DL1).
  Interventions: Drug: BNT323; Drug: BNT327
- Part 2 Cohort 1 - RP2D of BNT323 + BNT327 (Experimental)
  Interventions: Drug: BNT323; Drug: BNT327
- Part 2 Cohort 1 - Lower dose or RP2D of BNT323 + BNT327 (Experimental)
  Interventions: Drug: BNT323; Drug: BNT327
- Part 2 Cohort 1 - BNT323 monotherapy (Experimental): BNT323 monotherapy at a fixed dose
  Interventions: Drug: BNT323
- Part 2 Cohort 1 - BNT327 monotherapy (Experimental): BNT327 monotherapy at a fixed dose
  Interventions: Drug: BNT327
- Part 2 Cohort 2 - Selected dose level of BNT323 + BNT327 (Experimental)
  Interventions: Drug: BNT323; Drug: BNT327
- Part 2 Cohort 3 - Selected dose level of BNT323 + BNT327 (Experimental)
  Interventions: Drug: BNT323; Drug: BNT327
- Part 2 Cohort 4 - Selected dose level of BNT323 + BNT327 (Experimental)
  Interventions: Drug: BNT323; Drug: BNT327

INTERVENTIONS:
Drug: BNT323 — Intravenous infusion
  Arms: Part 2 Cohort 1 - BNT323 monotherapy; Part 2 Cohort 1 - Lower dose or RP2D of BNT323 + BNT327; Part 2 Cohort 1 - RP2D of BNT323 + BNT327; Part 2 Cohort 2 - Selected dose level of BNT323 + BNT327; Part 2 Cohort 3 - Selected dose level of BNT323 + BNT327; Part 2 Cohort 4 - Selected dose level of BNT323 + BNT327; Part1 - BNT323 + BNT327 combination therapy
Drug: BNT327 — Intravenous infusion
  Arms: Part 2 Cohort 1 - BNT327 monotherapy; Part 2 Cohort 1 - Lower dose or RP2D of BNT323 + BNT327; Part 2 Cohort 1 - RP2D of BNT323 + BNT327; Part 2 Cohort 2 - Selected dose level of BNT323 + BNT327; Part 2 Cohort 3 - Selected dose level of BNT323 + BNT327; Part 2 Cohort 4 - Selected dose level of BNT323 + BNT327; Part1 - BNT323 + BNT327 combination therapy

SUMMARY:
This is a Phase I/II, multi-site, open-label, two-part study designed to evaluate the efficacy, safety, optimized dose and contribution of components of BNT323 in combination with BNT327 in participants with hormone receptor-positive (HR+) or hormone receptor-negative (HR-), Human epidermal growth factor receptor (HER)2-positive, HER2-low (immunohistochemistry [IHC] 1+ or IHC 2+/in situ hybridization -), HER2-ultralow (IHC 0, with membrane staining) or HER2-null breast cancer (BC), or triple-negative breast cancer (TNBC).

DETAILED DESCRIPTION:
The study consists of two parts:

* Part 1 - Dose escalation: In this part of the study, participants with histologically confirmed, chemotherapy-pretreated advanced HR+, HER2-low or HER2-ultralow BC will receive BNT323 in combination with BNT327 (BNT323 + BNT327) in a dose escalation design. This will define the recommended Phase 2 dose (RP2D) for the BNT323 + BNT327 combination therapy.
* Part 2 - Dose optimization and exploratory cohorts: This part of the study will be an expansion phase, aiming to evaluate the efficacy and safety of the optimal dose combination and providing a more robust comparison against the other treatments. It will start once the enrollment in Part 1 is completed and the sponsor in conjunction with the Safety Review Committee has assessed available Part 1 efficacy and safety data. Part 2 of the study will have four cohorts, i.e., Cohorts 1 (dose optimization cohort), and Cohorts 2, 3, and 4 (exploratory cohorts). Recruitment to Cohorts 2, 3, and 4 will begin with RP2D from Part 1 and in parallel to randomization in Cohort 1.

Randomization is planned for Cohort 1 in Part 2, i.e., participants will be randomized in 2:2:1:1 ratio into one of the four arms (RP2D of BNT323 + BNT327, lower dose of RP2D of BNT323 + BNT327, BNT323 monotherapy, and BNT327 monotherapy). No randomization is planned for any other cohort in Part 2.

ELIGIBILITY:
Key Inclusion Criteria (applicable to all participants and all parts unless otherwise specified):

* Have pathologically documented BC that:

  * Is locally advanced, unresectable or metastatic.
  * Has a confirmed HER2 status as determined by the local laboratory (Part 1, Part 2 Cohorts 2 and 4) or the central laboratory (Part 2, Cohorts 1 and 3) from the most recently collected pre-randomization tumor sample.
  * Has a documented history of HER2 expression consistent with the subgroup definitions (i.e., HER2-low, HER2-ultralow, HER2-null, HER2-positive, or TNBC) as per current American Society of Clinical Oncology/College of American Pathologists guidelines.
* Have measurable disease defined by RECIST v1.1.
* Has left ventricular ejection fraction ≥55% by either echocardiography or multi-gated acquisition (scanning) within 28 days before randomization/enrollment.

Key Exclusion Criteria:

* Have history of small bowel obstruction requiring hospitalization within the past 3 months prior to the first dose of IMP.
* Have an uncontrolled intercurrent illness that would limit compliance with study requirement or substantially increase risk of incurring adverse events.
* Have clinically uncontrolled pleural effusion, ascites or pericardial effusion requiring drainage, peritoneal shunt, or cell-free concentrated ascites reinfusion therapy within 2 weeks prior to randomization/enrollment.
* Have a history of (non-infectious) interstitial lung disease (ILD)/pneumonitis that required steroids, have current ILD/pneumonitis, or where suspected ILD/pneumonitis cannot be ruled out by imaging at screening.
* Had prior treatment with topoisomerase I inhibitors, including ADCs with topoisomerase I inhibitor payloads such as trastuzumab deruxtecan.
* Have received any of the following therapies or drugs prior to the initiation of the study:

  * Participants who have previously been randomized to or received treatment in a previous study with BNT323, regardless of treatment assignment.
  * Participants who received prior treatment with a PD-L1/VEGF bispecific antibody. Note: Prior treatment with PD-1/VEGF bispecific antibodies, PD-1/PD-L1 inhibitors or anti-VEGF therapies are permitted.
  * Have received other systemic immunostimulatory agents or immunosuppressive therapies (such as interferon-α, interleukin-2, or methotrexate) within 4 weeks prior to the initiation of study treatment or are within five half-lives of the treatment drug (whichever is longer). Exception: excluding local, intranasal, intraocular, intra-articular or inhaled corticosteroids, short term use (≤7 days) of corticosteroids for prophylaxis (e.g., prevention of contrast agent allergy) or treatment of non-autoimmune conditions (e.g., delayed hypersensitivity reactions caused by exposure to allergens).
  * Have received systemic corticosteroids (at a dosage greater than 10 mg/day of prednisone or an equivalent dose of other corticosteroids) within 3 weeks prior to the initiation of study treatment.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 380 (Estimated)
Dates: Start 2025-04-23 (Actual); Primary Completion 2028-05 (Estimated); Study Completion 2029-05 (Estimated)

PRIMARY OUTCOMES:
Part 1 - Occurrence of dose limiting toxicities (DLTs) | During the DLT evaluation period (Cycle 1), i.e., the time of initiation of the first dose of investigational medicinal product (IMP) up to 21 days
  By dose level.
Occurrence of Treatment-emergent adverse events (TEAEs), Grade ≥3 TEAEs, serious adverse events (SAEs), treatment-related TEAEs, treatment-related Grade ≥3 TEAEs, and treatment-related SAEs | From the time of initiation of the first dose of IMP to 90 days after the last IMP dose
  In Part 1 by dose level. In Part 2 by cohort and arm.
Occurrence of dose interruption, reduction, and discontinuation due to TEAEs | From the time of initiation of the first dose of IMP to 90 days after the last IMP dose
  In Part 1 by dose level. In Part 2 by cohort and arm.
Part 2 - Objective response rate (ORR) | From the time of initiation of the first dose of IMP to last tumor assessment scan, i.e., up to 36 months.
  ORR defined as the proportion of participants in whom a confirmed complete response (CR) or partial response (PR) (per Response Evaluation Criteria in Solid Tumors version 1.1 [RECIST v1.1] based on the investigator's assessment) is observed as best overall response.
  By cohort and arm.

SECONDARY OUTCOMES:
Part 1 - ORR | From the time of initiation of the first dose of IMP to last tumor assessment scan, i.e., up to 36 months.
  ORR defined as the proportion of participants in whom a confirmed CR or PR (per RECIST v1.1 based on the investigator's assessment) is observed as best overall response.
  By dose level.
Part 2 - Duration of response (DoR) | From the time of initiation of the first dose of IMP to last tumor assessment scan, i.e., up to 36 months.
  DoR defined as the time from first objective response (CR or PR per RECIST v1.1 based on the investigator's assessment) to first occurrence of objective tumor progression (progressive disease [PD], per RECIST v1.1 based on the investigator's assessment) or death from any cause, whichever occurs first.
  By cohort and arm.
Part 2 - Disease control rate (DCR) | From the time of initiation of the first dose of IMP to last tumor assessment scan, i.e., up to 36 months.
  DCR defined as the proportion of participants with confirmed CR, PR, or stable disease (per RECIST v1.1 based on the investigator's assessment) as best overall response.
  By cohort and arm.
Part 2 - Time to response (TTR) | From the time of initiation of the first dose of IMP to last tumor assessment scan, i.e., up to 36 months.
  TTR defined as the time from first dose of IMP to first objective response (CR or PR per RECIST v1.1 based on the investigator's assessment).
  By cohort and arm.
Part 2 Cohort 1 only - Progression free survival (PFS) | From the time of initiation of the first dose of IMP to last tumor assessment scan, i.e., up to 36 months.
  PFS based on the investigator's assessment defined as the time from first dose of IMP to the first objective tumor progression (PD per RECIST v1.1) or death from any cause, whichever occurs first.
  By arm.

CONTACTS AND LOCATIONS:
Overall Officials: BioNTech Responsible Person, Study Director — BioNTech SE
Locations (18):
- United States (7):
  - Hematology - Oncology Associates of the Treasure Coast, Port Saint Lucie, Florida
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - START Midwest, LLC, Grand Rapids, Michigan
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Summit Medical Group, Florham Park, New Jersey
  - Memorial Sloan Kettering Hospital, New York, New York
  - South Texas Accelerated Research Therapeutics (START), LLC, San Antonio, Texas
- China (5):
  - Jilin Cancer Hospital, Changchun
  - Sichuan Cancer Hospital, Chengdu
  - Sichuan Provincial People's Hospital, Chengdu
  - Huizhou First Hospital, Huizhou
  - Fudan University Shanghai Cancer, Shanghai
- LLC Arensia Exploratory Medicine, Tbilisi, Georgia
- Institute of Oncology Arensia Exploratory Medicine, Chisinau, Moldova
- United Kingdom (4):
  - Addenbrooke s Hospital, Cambridge
  - Velindre Cancer Centre, Cardiff
  - St James's University Hospital, Leeds
  - Royal Free Hospital, London

IPD SHARING:
Plan to Share IPD: No